CLINICAL TRIAL: NCT04860778
Title: An Open-label, Exploratory Study to Investigate the Efficacy of BDNF Essentials® on Cognition in a Healthy Adult Population With Self-reported Memory Complaints
Brief Title: An Open-label, Exploratory Study to Investigate the Efficacy of BDNF Essentials® on Cognition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Researched Nutritionals LLC (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21BCHR
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Cognitive Change

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BDNF Essentials (Experimental): A proprietary blend of botanical extracts and isolates.
  Interventions: Dietary Supplement: BDNF Essentials

INTERVENTIONS:
Dietary Supplement: BDNF Essentials — Participants will take two capsules, twice daily with water for 84 days.

SUMMARY:
The objective of this open-label, exploratory study is to investigate the efficacy of BDNF Essentials® on cognition in a healthy adult population with self-reported memory complaints. As there is a dearth of available literature on BDNF in this study population, the current study is designed to understand the role of BDNF to inform potential future studies.

DETAILED DESCRIPTION:
The objective of this open-label, exploratory study is to investigate the efficacy of BDNF Essentials® on cognition in a healthy adult population with self-reported memory complaints. As there is a dearth of available literature on BDNF in this study population, the current study is designed to understand the role of BDNF to inform potential future studies. The study population represents a target group of individuals who would benefit from safe and efficacious nutraceuticals for the support of cognitive function. This transitional stage from normal cognition to cognitive impairment is viewed as an opportune window for intervention. This population of participants is being recruited to expand on previously published work on these individual ingredients while limiting confounding variables that could influence outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 45 years of age and older
* Waist circumference < 102 cm (40 inches) in men and < 88 cm (35 inches) in women
* Female participant is not of child-bearing potential, defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to enrollment

Or,

Females of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:

* Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
* Double-barrier method
* Intrauterine devices
* Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
* Vasectomy of partner at least 6 months prior to enrollment

  * A score of ≥ 24 on the Mini-Mental State Examination (MMSE 2)
  * Self-reported memory complaints as assessed by the revised Everyday Memory Questionnaire (EMQ) (with a score of ≥ 32)
  * Agrees to maintain current exercise routine, sleep and dietary patterns throughout the study
  * Agrees to avoid high caffeine consumption 24-hours prior to study appointments (examples include but not limited to no more than 2 cups of caffeinated coffee or tea)
  * Agrees to avoid alcohol consumption 24-hours prior to study appointments
  * Willingness to complete questionnaires, and diaries associated with the study and to complete all appointments
  * Provided voluntary, written, informed consent to participate in the study
  * Healthy as determined by medical history and laboratory results as assessed by the QI

Exclusion Criteria:

* Women who are pregnant, breast feeding, or planning to become pregnant during the study
* Allergy, sensitivity, or intolerance to the investigational product's active or inactive ingredients
* Dementia and/or cognitive decline or use of prescribed medications used to for dementia and/or cognitive decline (Section 6.3.1)
* Prescribed medications for depression that may affect concentration, attention and performance as assessed by the QI (Section 6.3.1)
* Current use of supplements used for cognition or mood support unless on a stable dose (Section 6.3.2)
* History of epilepsy, brain injury or trauma as assessed by the QI
* Self-reported confirmation of sleep disorder as assessed by the QI
* Prescribed or over-the-counter medications or supplements used for sleep (Section 6.3.1 and 6.3.2)
* Self reported colour-blindness
* Prescribed use of antibiotics within 1 month of baseline (Section 6.3.1)
* Prescribed use of anticoagulants/antiplatelets (Section 6.3.1)
* Prescribed or chronic use of over-the-counter anti-inflammatory medications (Section 6.3.1 and 6.3.2)
* Current use of supplements containing the ingredients in the IP unless willing to washout (Section 6.3.2)
* Current employment that calls for rotating shift work or shift work that will disrupt normal circadian rhythm in the last 3 weeks
* Travelled across 1 or more time zones in the last 3 weeks and/or is anticipating more travel during the study
* Use of medical cannabinoid products
* Current chronic use of cannabinoid products (>8 times/month) and is unwilling to stop for the duration of the study beginning 1 week prior to baseline. History of chronic use and occasional use to be assessed by QI on a case-by-case basis
* Use of tobacco, nicotine, or e-cigarette products within 12 weeks of baseline and during the study period
* Self-reported alcohol or drug abuse within the last 12 months
* Self-reported confirmation of HIV-, Hepatitis B- and/or C-positive diagnosis
* Autoimmune disease including Type I diabetes or are immune compromised
* Self-reported current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be assessed by the QI
* Clinically significant abnormal laboratory results at screening as assessed by the QI
* Blood donation 30 days prior to enrollment, during the study, or a planned donation within 30 days of the last study appointment
* Participation in other clinical research studies 30 days prior to enrollment will be assessed on a case-by-case basis by the QI
* Individuals who are unable to give informed consent
* Any other condition or lifestyle factor, that, in the opinion of the QI may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function | baseline to day 84
  Assessed using the Computerized Mental Performance Assessment System (COMPASS) test score for memory
Change in cognitive function | baseline to day 84
  Assessed using the Computerized Mental Performance Assessment System (COMPASS) test score for attention
Change in cognitive function | baseline to day 84
  Assessed using the Computerized Mental Performance Assessment System (COMPASS) test score for processing speed
Change in cognitive function | baseline to day 84
  Assessed by plasma Brain-Derived Neurotrophic Factor (BDNF) levels

SECONDARY OUTCOMES:
Change in plasma BDNF levels | baseline to day 28
  Assessed using the Computerized Mental Performance Assessment System (COMPASS)
Change in plasma BDNF levels | baseline to day 56
Change in memory | baseline to day 28
  Assessed using the Computerized Mental Performance Assessment System (COMPASS) test score for memory
Change in memory | baseline to day 56
  Assessed using the Computerized Mental Performance Assessment System (COMPASS) test score for memory
Change in attention | baseline to day 28
  Assessed using the Computerized Mental Performance Assessment System (COMPASS) test score for attention
Change in attention | baseline to day 56
  Assessed using the Computerized Mental Performance Assessment System (COMPASS) test score for attention
Change in processing speed | baseline to day 28
  Assessed using the Computerized Mental Performance Assessment System (COMPASS) test score for processing
Change in processing speed | baseline to day 56
  Assessed using the Computerized Mental Performance Assessment System (COMPASS) test score for processing
Change in mood | baseline to day 28
  Assessed by the Profile of Mood States (POMS) score
Change in mood | baseline to day 56
  Assessed by the Profile of Mood States (POMS) score
Change in mood | baseline to day 84
  Assessed by the Profile of Mood States (POMS) score
Change in Sleep | baseline to day 28
  Assessed by the Sleep Quality Questionnaire score
Change in Sleep | baseline to day 56
  Assessed by the Sleep Quality Questionnaire score
Change in Sleep | baseline to day 84
  Assessed by the Sleep Quality Questionnaire score
Change in Stress | baseline to day 28
  Assessed by the Perceived Stress Scale Score
Change in Stress | baseline to day 56
  Assessed by the Perceived Stress Scale Score
Change in Stress | baseline to day 84
  Assessed by the Perceived Stress Scale Score
Change in salivary cortisol levels | baseline to day 84
Change in serum Interleukin (IL-6) levels | baseline to day 84
Change in serum Tumour Necrosis Factor (TNF-alpha) levels | baseline to day 84

OTHER OUTCOMES:
Change in body weight | baseline to day 84
Incidence of adverse events | screening to day 84
Change in systolic blood pressure | baseline to day 84
Change in diastolic blood pressure | baseline to day 84
Change in heart rate | baseline to day 84
Change in aspartate aminotransferase (AST) | baseline to day 84
Change in alanine aminotransferase (ALT) | baseline to day 84
Change in alkaline phosphatase (ALP) | baseline to day 84
Change in total bilirubin | baseline to day 84
Change in creatinine | baseline to day 84
Change in sodium | baseline to day 84
Change in potassium | baseline to day 84
Change in chloride | baseline to day 84
Change in glucose | baseline to day 84
Change in estimated glomerular filtration rate (eGFR) | baseline to day 84
Change in neutrophil count | baseline to day 84
Change in eosinophil count | baseline to day 84
Change in basophil count | baseline to day 84
Change in lymphocyte count | baseline to day 84
Change in monocyte count | baseline to day 84
Change in red blood cell count | baseline to day 84
Change in hemoglobin | baseline to day 84
Change in hematocrit | baseline to day 84
Change in platelet count | baseline to day 84
Change in mean corpuscular volume | baseline to day 84
Change in mean corpuscular hemoglobin | baseline to day 84
Change in mean corpuscular hemoglobin concentration | baseline to day 84
Change in red cell distribution width | baseline to day 84

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, M.D., Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided